CLINICAL TRIAL: NCT06623409
Title: A Phase 1, Randomized, Double-Blind, Comparator-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of V540B in Healthy Adults.
Brief Title: Safety and Immunogenicity of V540B in Healthy Adults (V540B-002).
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: V540B-002; V540B-002 (Other: MSD)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GARDASIL®9 (G9) (Active Comparator): Participants will receive vaccinations with G9.
  Interventions: Biological: GARDASIL®9 (G9)
- V540B (Experimental): Participants will receive vaccinations with V540B.
  Interventions: Biological: V540B

INTERVENTIONS:
Biological: GARDASIL®9 (G9) — Suspension administered via intramuscular (IM) injection
  Other Names: V503
  Arms: GARDASIL®9 (G9)
Biological: V540B — Experimental vaccine and adjuvant administered via IM injection
  Arms: V540B

SUMMARY:
Researchers are looking for new ways to prevent cancers related to human papillomavirus (HPV). HPV is a common virus that can cause an infection. There are many different types of HPV. Most people's immune system can fight HPV infection and it goes away without treatment. For some people, HPV infections can last longer and may cause cancer years later.

A standard vaccine to prevent HPV-related cancers is GARDASIL®9 (G9). G9 protects against 9 types of HPV but it does not protect against other types of HPV. The study vaccine (called V540B) is designed to protect against the same HPV types that G9 protects against plus other HPV types. The main goal of this study is to learn about the safety of V540B in healthy adults and if people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health based on medical history, physical examination, vital sign (VS) measurements and electrocardiograms (ECGs) performed before randomization.

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of abnormal Pap smears, HPV- related external genital lesions (eg,condyloma acuminate, vulval intraepithelial neoplasia (VIN), or prostatic intraepithelial neoplasia (PIN)) or external genital cancer (eg, penile cancer), HPV-related vaginal or anal lesions (eg, condyloma acuminata or vaginal intraepithelial neoplasia (VaIN)) or vaginal or anal cancer.
* Has a history of cancer (malignancy).
* Has received any HPV vaccine or is expected to receive any HPV vaccine during the study, outside the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Solicited Injection-Site Adverse Event (AE) | Up to approximately 6 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Experience a Solicited Systemic AE | Up to approximately 6 months
  Solicited systemic AEs include headache, fatigue, nausea, dizziness, muscle aches, joint pain.
Immediate Reactions Occurring Within 30 Minutes After Any Vaccination | Up to approximately 6 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Experienced Unsolicited AEs | Up to approximately 7 months
  An unsolicited AE is an AE that was not solicited using a vaccine report card (VRC) and that is communicated by a participant (or their legally acceptable representative, if applicable). Unsolicited AEs include serious and nonserious AEs.
Number of Participants Who Experienced a Serious Adverse Event | Up to approximately 18 months
  Serious adverse events (SAEs) include adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
Number of Participants Who Experienced a Medically-Attended AE | Up to approximately 18 months
  AEs in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency department visit, office visit, or an urgent care visit with any medical personnel for any reason. Routine visits are not considered medically-attended adverse events (MAAEs). Examples of routine visits include physical examination, wellness visits, or vaccinations.
Number of Participants Who Experienced an Event of Clinical Interest | Up to approximately 18 months
  Events of clinical interest (ECIs) are defined as an overdose of Sponsor's product, drug-induced liver injury events, or potential immune-mediated diseases (pIMDs).

SECONDARY OUTCOMES:
Total Immunoglobulin G (IgG) Geometric Mean Ratios (GMRs) for anti-HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | Up to approximately 7 months
  Geometric mean ratio (GMR) of titers for participants vaccinated with V540B versus those who received G9 alone will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (5):
  - Anaheim Clinical Trials ( Site 0002), Anaheim, California
  - California Clinical Trials Medical Group managed by PAREXEL ( Site 0008), Glendale, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0003), Hallandale, Florida
  - Research Centers of America ( Hollywood ) ( Site 0001), Hollywood, Florida
  - Velocity Clinical Research, Omaha ( Site 0005), Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com